CLINICAL TRIAL: NCT04420819
Title: Effects of Ischemic Preconditioning on Muscle Damage Induced by Excentric Exercise: Randomized Clinical Trial Placebo Controlled
Brief Title: Effects of Ischemic Preconditioning on Muscle Damage Induced by Excentric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal Investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FCT/UNESP
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Ischemic Preconditioning; Exercise; Musculoskeletal Pain; Creatine Kinase; Muscle Fatigue; Stress, Physiological
MeSH Terms: conditions — Motor Activity; Musculoskeletal Pain | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IPC-LOP (Experimental): this group will carry out the baseline assessments, perform the ischemic preconditioning using exactly the limb occlusion pressure , then perform post-IPC assessments and start the excentric exercise, and the post-exercise assessments will take place immediately after the end of the EE and will be repeated in 24h, 48h, 72h and 96h.
  Interventions: Device: Ischemic Preconditioning
- IPC-40% (Experimental): this group will carry out baseline assessments, perform IPC using 40% more occlusion than LOP, then perform assessments after IPC protocol and start EE, and post exercise assessments will take place immediately after the end of EE and will be repeated in 24h, 48h, 72h and 96h.
  Interventions: Device: Ischemic Preconditioning
- IPC-10mmHg: (Placebo Comparator): this group will perform baseline assessments, perform occlusion-perfusion intervention with 10 mmHg restriction characterizing the placebo, then perform post-IPC assessments and initiate EE, and post-exercise assessments will take place immediately after completion of EE and if will repeat in 24h, 48h, 72h and 96h.
  Interventions: Device: Ischemic Preconditioning
- CONTR (No Intervention): this group will carry out the baseline assessments, immediately after starting the EE, and the post-exercise assessments will happen immediately after the end of the EE and will be repeated in 24h, 48h, 72h and 96h.

INTERVENTIONS:
Device: Ischemic Preconditioning — The IPC is characterized by the application of brief periods of circulatory occlusion (ischemia) and reperfusion of a limb in the minutes to hours that precede the exercise through the insufflations and deflations of a pressure cuff
  Arms: IPC-10mmHg:; IPC-40%; IPC-LOP

SUMMARY:
Introduction: eccentric exercise (EE) has been widely used in rehabilitation and in improving physical fitness due to its mechanical advantage and less metabolic demand, however, EE can induce muscle damage providing structural changes and reduced muscle function, therefore, it is necessary to look for alternatives to reduce this damage caused by stress. Thus, ischemic preconditioning (PCI) can be seen as an aid in reducing the damage caused by EE, as it can attenuate the ischemia-reperfusion injury, and can be used to accelerate the post-exercise recovery process. Objectives: to compare the effects of PCI, using different occlusion pressures, on acute and late responses to perceptual outcomes and muscle injury markers, in addition to checking whether the technique causes deleterious effects on performance in post-exercise recovery. Methods: a randomized placebo controlled clinical trial will be conducted with 80 healthy men aged 18 to 35 years who will be randomly divided into four groups: PCI using total occlusion pressure (POT), PCI with 40% more than POT, placebo (10 mmHg) and control. The PCI protocol will consist of four cycles of ischemia and reperfusion of five minutes each. All groups will perform an EE protocol, initial assessments, immediately after the end of the EE, 24, 48, 72 and 96 hours after exercise, with the maximum isometric voluntary contraction (CVIM) assessed by the isokinetic dynamometer, vectors of cell integrity by by means of electrical bioimpedance (BIA), creatine kinase (CK), blood lactate, pain on the visual analog scale (VAS), pain threshold by the pressure algometer, and tone, muscle rigidity and elasticity by myotonometry. The descriptive statistical method and analysis of variance will be used for the repeated measures model. The level of significance will be p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* not having any health condition that contraindicates or prevents EE;
* not having diagnosed diabetes and high blood pressure;
* not having inflammatory, psychiatric, cardiovascular and / or respiratory rheumatic disease;
* not being an alcoholic, using drugs and / or a smoker;
* without a history of knee surgery (for example, meniscal repair and ligament reconstruction) or recent musculoskeletal injury to the lower limbs that may impair performance during tests or interventions (for example, muscle injury, tendinopathy, patellofemoral pain in the lower limbs and / or back pain in the last six months);
* without involvement in any type of training program during the study period;
* not being engaged in the lower limb strength training program during the three months prior to participating in the study;
* not using ergogenic supplements to improve physical performance and / or muscle mass and / or vasoactive drugs;
* not having one or more risk factors predisposing to thromboembolism.

Exclusion Criteria:

* present a health problem that does not allow continuity,
* use medication, electrotherapy or other therapeutic means that may interfere with any result;
* perform unusual or strenuous physical activities during the evaluation period;
* want to leave the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Muscle damage | Change from baseline at 96 hours after exercise
  Plasma CK concentration will be obtained by means of 32 μL of capillary blood collected from the digital pulp.
Blood lactate concentration | Change from baseline at 96 hours after exercise
  Blood lactate concentration of the participant will be collected 25 ml of blood with an ear lobe capillary
Muscle strength in isokinetic | Change from baseline at 96 hours after exercise
  Maximal voluntary isometric contraction (MVIC)

SECONDARY OUTCOMES:
Muscle pain | Change from baseline at 96 hours after exercise
  Assessed using a visual analog scale that ranges from 0 to 10 points, the higher the score, the worse the result.
Pain threshold | Change from baseline at 96 hours after exercise
  Assessed using pressure algometer equipment, and the pain threshold will be classified according to the cut-off point of 2.55kgf. Participants will be classified as "sensitive to pain" if they have values below 2.55kgf.
Resistance through Bioimpedance analysis (BIA) | Change from baseline at 96 hours after exercise
  Evaluation of tissue resistance, the higher the value, the worse the result
Reactance through Bioimpedance analysis (BIA) | Change from baseline at 96 hours after exercise
  Evaluation of tissue reactance, the higher the value, the better the cell integrity
Phase angle through Bioimpedance analysis (BIA) | Change from baseline at 96 hours after exercise
  Assessment of the phase angle, the higher the value, the better the condition of the participant
Tone muscular through Myotonometry used the MyotonPRO equipment | Change from baseline at 96 hours after exercise
  Natural Oscillation Frequency [Hz], characterizing Tone of the quadriceps femoris muscle
Stiffness through Myotonometry used the MyotonPRO equipment | Change from baseline at 96 hours after exercise
  Dynamic Stiffness [N/m] of the quadriceps femoris muscle
Elasticity through Myotonometry used the MyotonPRO equipment | Change from baseline at 96 hours after exercise
  Mechanical Stress Relaxation Time [ms] featuring muscle elasticity of the quadriceps femoris muscle
Perception of recovery | Change from baseline at 96 hours after exercise
  Perception of recovery was obtained using a 10-point Likert Scale, with a rating of 1 indicating the feeling "not recovered" and a rating of 10 the feeling "fully recovered"

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pizzo Junior E, de Souza Cavina AP, Lemos LK, Biral TM, Pastre CM, Vanderlei FM. Effects of different ischemic preconditioning occlusion pressures on muscle damage induced by eccentric exercise: a study protocol for a randomized controlled placebo clinical trial. Trials. 2021 May 5;22(1):326. doi: 10.1186/s13063-021-05285-7. PMID 33952329